CLINICAL TRIAL: NCT03146104
Title: Comparison of Total Intravenous Anesthesia vs. Inhalational Anesthesia on Brain Relaxation, Subdural Pressure and Hemodynamics in Patients With Acute Subdural Hematoma Undergoing Emergency Craniotomy- A Randomized Control Trial
Brief Title: Comparison of Total Intravenous Anesthesia vs. Inhalational Anesthesia in Acute Subdural Hematoma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr.Preethi.J, Principal investigator, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PGRMC-27.10.2016/29
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Acute Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Acute | interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Active Comparator): Maintenance of anesthesia with 100-150mcg/kg/min propofol, O2 and air and FiO2 of 40%
  Interventions: Drug: Propofol
- Group I (Active Comparator): Maintenance of anesthesia with 1 MAC of isoflurane,O2 and air and FiO2 of 40%
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Propofol — Intraoperative anesthesia will be maintained using propofol 100-150 mcg/kg/min, oxygen and air and FiO2 of 40% in propofol group (GROUP P)
  Arms: Group P
Drug: Isoflurane — in(GROUP I) maintenance will be done with 1 MAC of isoflurane, oxygen and air and FiO2 of 40%.
  Arms: Group I

SUMMARY:
Consent will be taken from the relatives and the patient will be taken to the operating room. Inside the operation theatre patient will be shifted to operating table and standard monitors will be attached. The patient will then be given induction agent to make him/her unconscious and unaware of the surrounding and muscle relaxant to prevent movement will be administered. He/she will be intubated with appropriate size tube to maintain airway. In order to maintain anesthesia he/ she will be given either of inhalational or intravenous anesthetic throughout the surgery. Intracranial pressure will be measured using venflon needle as soon as burr hole is created in the skull. Throughout the surgery patients vital parameters will be monitored and appropriate treatment will be given in case if the vitals are not stable.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be enrolled in the study and randomized into one of the two group's propofol - P and isoflurane - I. Preoperative Glasgow coma scale (GCS) and computer tomography (CT) findings will be recorded. Intraoperatively peripheral intravenous line will be secured, standard monitors including non invasive blood pressure (NIBP), electrocardiogram (ECG), heart rate (HR), pulse oximetry, SPO2 probe will be connected. Pre-oxygenation will be done with 100% O2 for 3 minutes. In both the groups induction will be done using 3 mcg/kg fentanyl, 2 mg/kg propofol and muscle relaxation will be achieved with 0.1mg/kg vecuronium. Post induction patients will be intubated with appropriate size endotracheal tube (male with 8.0 and female with 7.0) and radial artery will be cannulated with zero pressure adjustment at mid axillary line for continuous blood pressure monitoring and blood sampling. Central line will be secured using 7 French triple lumen central venous catheter in the subclavian vein or internal jugular vein. Cardiac output monitor (EV1000) will be connected to arterial and central line and values of stroke volume (SV), systemic vascular resistance (SVR), cardiac output (CO) and cardiac index (CI) will be obtained. Intraoperative anesthesia will be maintained using propofol 100-150 mcg/kg/min, oxygen and air and FiO2 of 40% in propofol group (GROUP P) whereas in isoflurane group (GROUP I) maintenance will be done with 1 MAC of isoflurane, oxygen and air and FiO2 of 40%. In both the groups Etco2 will be maintained at 32-33 mmHg. HR and IBP will be kept within +/- 20% of the baseline values. If the systolic blood pressure decreases more 20% of base line, crystalloids will be given as initial management and failing to improve blood pressure, vasopressors namely phenylephrine or dopamine will be given intravenously. At the time of scalp incision mannitol 1 gm/kg will be given over 20min. On creating first burr hole a 22G/0.8mm venflon cannula will be placed under dura and connected to a pressure transducer system via a polyethylene catheter. Zero level of ICP will be adjusted with the transducer kept at the level of mastoid process(6). The pressure measured will be the estimate for intracranial pressure. Cerebral perfusion pressure (CPP) will be calculated as the difference between mean arterial pressure MAP and ICP. If the intracranial pressure is more than 25 mmHg then moderate hyperventilation will be given with Etco2 of 25-28 mmHg. Once the dura is opened brain relaxation score will be assessed on four point scale, using tactile evaluation by neurosurgeon who will be blinded to anaesthetic technique. The tension will be categorized as follows:

1. Perfectly relaxed
2. Satisfactorily relaxed
3. Firm brain
4. Bulging brain Meanwhile hemodynamic stability in terms of heart rate, blood pressure, MAP, cardiac output, stroke volume , stroke volume variation, systemic vascular resistance, cardiac index, and cerebral perfusion pressure will be measured before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes until surgery is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients posted for emergency craniotomy with TBI having

  * Subdural hematoma
  * GCS < 8
  * Age 18 to 60 years.
  * Both males and females

Exclusion Criteria:

* Extradural hematoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Brain relaxation score | At the time of dura opening

SECONDARY OUTCOMES:
intracranial pressure | at the time of creating first burr hole
blood pressure | Before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
Mean arterial pressure | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
heart rate | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
Cardiac output | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
Stroke volume | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
Stroke volume variations | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
systemic vascular resistance | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
cardiac index | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours
cerebral perfusion pressure | before induction, at the time of induction and at 1 , 2, 3, 4, 5th minute after induction and thereafter every 15 minutes for a maximum of 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Preethi.J, Puducherry, India

REFERENCES:
- [Derived] Preethi J, Bidkar PU, Cherian A, Dey A, Srinivasan S, Adinarayanan S, Ramesh AS. Comparison of total intravenous anesthesia vs. inhalational anesthesia on brain relaxation, intracranial pressure, and hemodynamics in patients with acute subdural hematoma undergoing emergency craniotomy: a randomized control trial. Eur J Trauma Emerg Surg. 2021 Jun;47(3):831-837. doi: 10.1007/s00068-019-01249-4. Epub 2019 Oct 29. PMID 31664468